CLINICAL TRIAL: NCT03541837
Title: Ultrasound Guided Thoracic Erector Spinae Plane Blocks Within an Enhanced Recovery Program Decreases Opioids Consumption and Improves Patient Postoperative Rehabilitation After Open Cardiac Surgery: A Controlled Before-After Study
Brief Title: Erector Spinae Plane Block and Pain Management in Cardiac Surgery
Acronym: ESPCATHEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VINMEC HS
Record Dates: First submitted 2018-03-12; First posted 2018-05-31 (Actual); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Cardiac Surgery; Adult
Keywords: Bilateral ESP Catheter; Open heart surgery; opioid free post op analgesia
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Prospective series case compared to a before group of consecutive patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- peri operative analgesia (Other): Post operative regional analgesia by Erector Spinae bilateral catheters with infusion of ropivacaine
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — ESP catheter
  Other Names: ESP catheter

SUMMARY:
Evaluation of the benefit effects of Peri-Operative analgesia by Continuous Bilateral Erector Spinae Plane block(ESP) for Open Cardiac Surgery: A case series prospective study with a comparison a retrospective case series (Before and after)

DETAILED DESCRIPTION:
After Patient's information and consent from the Ethical committee of VinMec Healthcare (#06/2017/HDD-VMEC) the anesthesia team will perform to all adult patients for open heart surgery after the anesthesia induction a bilateral insertion of an Erector Spinae Plane Block catheter under ultrasound guidance The Block performance :

Patient in right lateral decubitus. The anesthesiologist will use an high-frequency linear ultrasound transducer sagitally at T4 level to identify the lateral extremity of the T4 transverse process (Logic E GE USE). After inserting in plane a Tuohy needle 80 mm 18G the anesthesiologist will locate the tip of the needle and confirm by hydrodissection the inter-fascial space between the inter-transverse ligament anteriorly and the fascia of the Erector Spinae Muscle posteriorly . He will insert under ultrasound vision a catheter (Perifix B.Braun Germany) . The anesthesiologist check the right position of the catheter with a dextrose 5% injection = 2mL under ultrasound vision and see the spread of the Dextrose between in the inter-fascial space. This procedure will be bilateral. The catheter will have a yellow label on the Huer®-Lock connector to identify clearly that it is regional analgesia catheter to prevent any errors in these patients will a lot of catheters.

After this control an induction dose of Ropivacaine (0.5%) 0.25mL/Kg is injected in each catheter ( Loading dose).

8 h after a automatic infusion of Ropivacaine (0.2%) will be infused throw the 2 ESP catheters the infusion regimen will be Intermittent automatic bolus every 6h. on each catheter. The bolus on the second catheter will be delayed by 1 hour to minor the maximal plasmatic concentration.

Volume of the bolus:

For 40 to 50 kg patient the volume of intermittent automatic bolus will be 6 mL/ 6H/ Side For 50 to 60 kg patient the volume of intermittent automatic bolus will be 8 mL / 6H/ Side For 60 to 70 kg patient the volume of intermittent automatic bolus will be 10 mL / 6H/ Side For a 70 kg and > 1.70 m Patient the volume of intermittent automatic bolus will be 12 mL / 6H/ Side

If the block extension is not enough additional bolus by clinician only of 8 mL maximum 3 per day and 1 hour after the last automatic bolus delivered

If the analgesia is not efficient after 1 additional bolus the catheters will be removed and we will prescribe the classical IV analgesia as before.

The regional analgesia will be up to 4 hours after mediastinal drain removal and a maximum of 76h. after catheter incision

A Bi Daily inspection of the catheters insertion points will be done. If redness around puncture point the catheters will be removed and shift to classical IV analgesia to prevent any infection.

The criteria studied will be:

Consumption of opioids at 48h Variation of Blood pressure during sternotomy Level of pain at rest and mob after the surgery Time to extubate the patient Early mobilisation after surgery the quality of thorax expansion Level of pain 1 month after the surgery and limited activity at one month

The control group was an historical group of twenty consecutive patients, operated by the same surgeons from June 8th 2017 and August 1th 2017 and matched with the studied group, in which data were noted just before the introduction of ESB in the ERAS program. All data from the control group come from the centralized computer network of patient records at Vinmec University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Consent signed
* Open heart surgery
* Hemodynamic stable after anesthesia induction No variation more than 20% of blood pressure

Exclusion Criteria:

* refusal by patient
* Unstable hemodynamic after induction
* Failure of ESP catheter insertion Must have 2 ESP catheter well inserted

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-02-25 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Post operative Opioids consumption | 48h.
  Total dose of morphine used in post operative in mg of Morphine

SECONDARY OUTCOMES:
Acute post op pain | 1 hour after extubation
  VAS Visual analogically scale from 0 to 10 at rest and Thorax mobilisation
Pain at one month after surgery | One month exactly = 30 days after date of surgery
  VAS Visual analogically scale from 0 to 10 at rest and mobilisation
Peri operative sufentanil consumption | from induction anesthesia to last point of the skin (end of surgery) Time unit Hour
  Total dose of sufentanil in msg/kg

CONTACTS AND LOCATIONS:
Overall Officials: huyen vu, Study Chair — VINMEC
Locations (1):
- VinMec Central park International hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
excel sheet
Supporting Information: Study Protocol, ICF, CSR
Time Frame: April for 2 months
Access Criteria: Director of research